CLINICAL TRIAL: NCT00700830
Title: Assessment of Safety and Efficacy of Levemir® (Insulin Detemir) Treatment for Insulin Naive Patients With Type 2 Diabetes Mellitus
Brief Title: Observational Study to Evaluate the Safety and Efficacy of Levemir® in Type 2 Diabetes
Acronym: IDEALS
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-3571
Record Dates: First submitted 2008-06-18; First posted 2008-06-19 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2013-12

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: insulin detemir

INTERVENTIONS:
Drug: insulin detemir — Initial dosage and the following dosages will be prescribed by the physician as a result of a normal clinical evaluation
  Other Names: Levemir®

SUMMARY:
This study is conducted in Africa. The aim of this study is to assess the safety and efficacy of Levemir® treatment for insulin naive patients with type 2 diabetes under normal clinical practice conditions in Algeria.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities
* Type 2 diabetes
* HbA1c between 7-9%
* Insulin naive
* Inadequate control with oral antidiabetics therapy as judged by investigator

Exclusion Criteria:

* Patients with type 1 diabetes
* Hypersensitivity to Levemir® or to any of the excipients
* Pregnancy, or desire of pregnancy within next 6 months
* HbA1c greater than or equal to 9%
* Known or suspected allergy to the trial product or to any of the excipients
* Subjects who are unlikely to comply with protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Type 2 diabetes insulin naive patients
Sampling Method: Non-Probability Sample
Enrollment: 1976 (Actual)
Dates: Start 2008-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Assessment the incidence of the Serious Adverse Events including the major Hypoglycaemia. | During study

SECONDARY OUTCOMES:
HbA1c | after 12 weeks (3 months) AND after 24 weeks (6 months)
FBG (Fasting Blood Glucose) | Monthly average for each month, and average of the past quarter
Weight | after 12 weeks (3 months) AND after 24 weeks (6 months)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Algiers, Algeria

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com